CLINICAL TRIAL: NCT00003223
Title: A Single Arm, Phase II Study to Determine the Safety and Efficacy of 4-HPRN-(4-Hydroxyphenyl) Retinamide for Treating Oral Intraepithelial Neoplasia
Brief Title: SWOG-9507, Fenretinide in Treating Patients With Neoplasia of the Mouth
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to poor accrual.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000066085; SWOG-9507 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-09-10 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
Keywords: lip and oral cavity cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms | interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): Fenretinide 200 mg PO days 1-25, q 28 days x 6 cycles.
  Interventions: Drug: fenretinide

INTERVENTIONS:
Drug: fenretinide — 200 mg/day PO, days 1-25 q 28 days x 6 cycles.
  Other Names: N-(4-hydroxyphenyl)retinamide, 4-HPR

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of fenretinide may be an effective way to prevent the development of cancer in patients with neoplasia of the mouth.

PURPOSE: Phase II trial to study the effectiveness of fenretinide in preventing cancer in patients who have neoplasia of the mouth.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of fenretinide in patients with oral intraepithelial neoplasia. II. Assess the toxicity of fenretinide in these patients.

OUTLINE: Patients receive oral fenretinide on days 1-25 every 28 days for a maximum of 6 courses. After 6 courses, patients receive a post-treatment biopsy. Patients exhibiting disease progression or unacceptable toxicities are removed from the study. Patients are followed at 3 and 6 months.

PROJECTED ACCRUAL: A total of 51 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven oral mucosal intraepithelial neoplasia Stage II: moderate dysplasia, keratosis with atypia Stage III: severe keratinizing or nonkeratinizing dysplasia No myelodysplastic syndrome No retinopathies

PATIENT CHARACTERISTICS: See General Eligibility Criteria

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No concurrent chemotherapy Endocrine therapy: No concurrent endocrine therapy Radiotherapy: No concurrent radiotherapy Surgery: Prior surgical ablation of prior dysplastic sites allowed Other: At least 2 months since prior therapy toxicities Patient Characteristics-- Age: Not specified Performance Status: SWOG 0-1 Life Expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception at least 1 month before, during, and at least 2 months after study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1997-12; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (15):
- United States (15):
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Kansas Medical Center, Kansas City, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah